CLINICAL TRIAL: NCT05924035
Title: Effect of Hyperbaric Oxygen Treatment (HBOT) on Recovery From Exercise
Brief Title: HBOT and Exercise Recovery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Needed additional support.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000035148
Record Dates: First submitted 2023-06-15; First posted 2023-06-29 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Exercise Recovery
Keywords: Hyperbaric Oxygen Treatment; Exercise Recovery; High Performance Athletes

STUDY DESIGN:
Intervention Model Description: The study is a prospective, case-controlled pilot study, performed over three weeks with 6 participants in each group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Group (No Intervention): Control Group will participate in standardized, prescribed exercise 4 days per week and perform countermovement jumps on a force plate both before and after daily workouts (standard of care summer athletic training)
- HBOT Treatment (Experimental): HBOT Treatment Group will receive HBOT Treatment in addition to standardized, prescribed exercise 4 days per week and perform countermovement jumps on a force plate both before and after daily workouts (standard of care summer athletic training)
  Interventions: Device: HBOT

INTERVENTIONS:
Device: HBOT — HBOT treatment on a multiplace chamber (OXYHeal Hyperbaric Oxygen Chamber), 100% oxygen at 2.0 atmospheres for 90 minutes - on 4 consecutive days within 3 hours of completion of exercise training (as soon as practically possible). This will occur during week 2 of data collection.
  Arms: HBOT Treatment

SUMMARY:
The purpose of this pilot study is to investigate the effect of hyperbaric oxygen treatment on recovery from exercise in high performance athletes. Outcome measures will be both physical outcome measures from a force plate, as well as physiologic measures of recovery (including blood lactate and muscle oxygenation) and perceived rates of exertion and recovery.

DETAILED DESCRIPTION:
Initial visit to discuss the study and obtain consent. At this visit, baseline subject demographics (height, weight, body composition) and a medical history will be taken to confirm that there are no medical contraindications to either exercise or HBOT. This visit will likely take 30-45 minutes.

There will be 15 subsequent visits. Each of these visits will be conducted concurrent with their standard off-season workouts. An additional 15 minutes per workout session may be required for the collection of study-related, non-standard of care, outcome measures.

During the second week of the study, the experimental group will have four daily 90 minute sessions of HBOT. Travel time from the site of their workouts (West Haven CT) to the HBOT facility (Bridgeport Hospital) is approximately 20 minutes.

Immediately following exercise, each experimental subject will be fitted with the surface muscle oxygenation monitor on their vastus lateralis. This monitor (Moxy, Fortiori Design LLC) utilizes near-infrared spectroscopy. The monitor will be applied to the distal third of the vastus lateralis muscle (12cm above the knee joint) as identified and marked by the PI (an orthopaedic surgeon). This will provide continuous muscle oxygenation report following exercise, including during and immediately after the HBOT treatment.

Both the experimental and control groups will have blood lactate measurements taken within 15 minutes before the start of their daily exercise, as well as within 5 minutes of the completion of exercise, utilizing The Edge blood lactate monitoring system (Apexbio, Taiwan). Once per week the performance of The Edge monitor will be validated utilizing The Edge Lactate Control Solution.

The Edge monitor measures blood lactate from a drop of blood from a finger tip applied to a sterile lancet. The result is reported in approximately 45 seconds.

ELIGIBILITY:
Inclusion Criteria:

* Yale University varsity student-athletes
* Cleared for unrestricted participation in varsity athletics training at the time of data collection
* No implantable electronic medical device (ie. Deep brain stimulator or insulin pump) or with other contraindication to HBOT
* Those who consent to participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2023-07 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Relative Peak Propulsive Power | within 3 hours of exercise completion during week 2
  Relative Peak Propulsive Power will be assessed as the peak instantaneous mechanical power applied to the system center of mass during the population phase relative to the system mass from a countermovement jump using the Hawkin Dynamic force plates.
modified Relative Strength Index (mRSI) | within 3 hours of exercise completion during week 2
  mRSI assessed as jump height calculated using the vertical velocity of the system center of mass at the instant of take-off divided by the total time taken from the initiation of movement to the instant of take-off using the Hawkin Dynamic force plates.
Average Landing Force | within 3 hours of exercise completion during week 2
  Average Landing Force assessed as the average vertical ground reaction force applied to the system center of mass during the landing phase using the Hawkin Dynamic force plates.

SECONDARY OUTCOMES:
Change in Muscle oxygenation | baseline and week 2
  Muscle oxygenation will be measured during and post exercise, with and without HBOT using a surface muscle oxygenation monitor on their vastus lateralis.
Change in Blood lactate | baseline and week 2
  Blood lactate will be measured pre- and post-exercises, and post-HBOT using The Edge blood lactate monitoring system. The Edge monitor measures blood lactate from a drop of blood from a finger tip applied to a sterile lancet. The result is reported in approximately 45 seconds.
Rate of Perceived Exertion (RPE) scale | daily up to 3 weeks
  The scale allows participants to subjectively rate their perceived level of exertion during exercise. It is scored from 0 (Nothing at all) to 11 (very, very hard) and reported using self-report. A higher score indicates more perceived exertion.
Rate of Perceived Recovery (RPR) scale | daily up to 3 weeks
  The scale allows participants to subjectively rate their perceived level of recovery from last exercise session. It is scored from 0 (very poor recovery/extremely tired) to 11 (very good recovery/extremely well-disposed) and reported using self-report. A higher score indicates more perceived recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Gardner, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes